CLINICAL TRIAL: NCT00034333
Title: Study of Doxorubicin Hydrochloride Adsorbed to Magnetic Targeted Carriers (MTC-DOX) Administered by Intrahepatic Delivery Versus Intravenous Doxorubicin for Treatment of Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Doxorubicin Adsorbed to Magnetic Beads Vs. IV Doxorubicin in Treating Liver Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: FeRx (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTC-DOX-004; NCT00052819 (obsolete NCT alias)
Record Dates: First submitted 2002-04-25; First posted 2002-04-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatoma; Unresectable adult primary liver cancer; liver cancer; HCC; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Injections

INTERVENTIONS:
Drug: MTC-DOX for Injection

SUMMARY:
MTC-DOX is Doxorubicin or DOX, a chemotherapy drug, that is adsorbed, or made to "stick", to magnetic beads (MTCs). MTCs are tiny, microscopic particles of iron and carbon. When DOX is added to MTCs, DOX attaches to the carbon part of the MTCs. MTC-DOX is directed to and deposited in the area of a tumor, where it is thought that it then "leaks" through the blood vessel walls. Once in the surrounding tissues, it is thought that Doxorubicin becomes "free from" the magnetic beads and will then be able to act against the tumor cells. The iron component of the particle has magnetic properties, making it possible to direct MTC-DOX to specific tumor sites in the liver by placing a magnet on the body surface. It is hoped that MTC-DOX used with the magnet may target the chemotherapy directly to liver tumors and provide a treatment to patients with liver cancer.

To be sure of the effect of MTC-DOX on liver cancer, it will be compared to the effect of Doxorubicin given through the vein.

The study treatments will be administered every three weeks, (which is considered a study treatment cycle), until you complete six treatment cycles, the tumor grows, disappears, or you experience a side effect, which may cause you to leave the study. Follow-up visits will occur on Days 3, 10, and 21 following treatment in the first cycle and Days 7 and 21 for the remaining cycles, and also 60 days after you receive your last treatment cycle.

Therefore, the purpose of this Phase 2/3 study is to evaluate safety, tolerance, and efficacy (survival time) of an MTC-DOX dosing strategy where the DOX dose is determined by tumor size

ELIGIBILITY:
Patients may be enrolled into this protocol only if all of the following inclusion criteria are met:

* Unresectable hepatocellular carcinoma diagnosed by CT scan and meets the criteria described in Section 23.
* Total combined cross-sectional area of all hepatic tumors as determined by CT scan is between 4 and 200 cm2.
* Center of the tumor(s) mass must be </= 14 cm from the anterior lateral abdominal wall as determined by cross-sectional imaging at baseline. This is required for optimal placement of the magnet. If more than one tumor mass is present, all of the tumor masses must meet this criterion.
* Is ambulatory with a Karnofsky performance status score > 60 and an estimated life expectancy of > 3 months.
* Is judged by the investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to allow follow-up.
* Have the ability to give informed written consent prior to initiation of therapy.
* If female and of childbearing potential,must have a negative beta-HCG prior to receiving treatment.
* Must agree to use an effective method of contraception

Patients will be excluded from enrollment if any of the following apply:

* Has a history of cancer other than hepatocellular (excluding resected basal cell carcinoma; or curatively resected stage 1 or less cervical cancer if disease free for 5 years or more).
* Has had prior local radiation therapy within the last 4 weeks, mediastinal radiation therapy within the last 3 months, or chemotherapy within the last 4 weeks.
* Diffuse hepatocellular carcinoma or disease that precludes delivery of the drug to the tumor via a vessel that feeds the tumor.
* Has another active medical condition(s) or organ disease(s) that may either compromise patient safety or interfere with the safety and/or outcome (e.g., survival) evaluation of the study drugs. While this exclusion is not limited to the following abnormalities, if any of the following laboratory abnormalities are present, the patient should be excluded:

WBC < 2,000 /uL Platelets < 50,000/uL Hemoglobin < 8.0 gm/dL Total bilirubin > 3.0 mg/dL ALT or AST >/= 5 x upper limit of normal Serum Creatinine >2.0 mg/dL INR >/= 1.5

* Has cardiac dysfunction with a left ventricular ejection fraction < 40%.
* Has clinically significant pulmonary impairment
* Plans concomitant chemotherapy, radiation therapy, hormonal and/or biological treatment for cancer including immunotherapy while on study.
* Has an indwelling cardiac pacemaker, cerebral aneurysm clips, or any other indwelling device or appliance that could be adversely affected by the use of the external magnet.
* Has documented evidence of hemachromatosis or hemosiderosis.
* Has CT or ultrasound evidence of portal vein invasion or thrombosis.
* Prior orthotopic hepatic transplant.
* Has received previous treatment with doxorubicin, idarubicin, and/or other anthracyclines or anthracenes.
* Has a known allergy to doxorubicin, MTC-DOX or any of their components.
* Has been treated with any investigational drug, investigational biologic, or investigational therapeutic device within 30 days of initiating study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Joy Koda, Ph.D., Study Chair — FeRx
Locations (29):
- United States (11):
  - Long Beach VA Medical Center, Long Beach, California
  - VAMC San Francisco and Comprehensive Cancer Ctr., San Francisco, California
  - Northwestern Univ. Med. School, Chicago, Illinois
  - Weill Medical College of Cornell University, New York, New York
  - Univ. of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Scott & White Mem. Hosp. & Clinic, Temple, Texas
  - McGuire DVAMC, Richmond, Virginia
- Austria (2):
  - Landeskrankenhaus Graz University Hospital, Graz
  - University Hospital Vienna, Vienna
- Germany (2):
  - University Hospital Cologne, Cologne
  - University Hospital Am Main, Frankfurt
- Hong Kong (2):
  - Queen Mary Hospital, University of Hong Kong, Pokfulam
  - Chinese Universtiy of Hong Kong, Shatin, N.T.
- Russia (2):
  - Central Research Institute of Roentgenology and Radiology, Pesochny, Sankt-Peterburg
  - N.N. Blokhin Cancer Research Center RAMS, Moscow
- Thailand (5):
  - Chulalongkorn University Hospital, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - National Cancer Institute, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen Universtiy, Khon Kaen
- Institute of Oncology AMS of Ukraine, Kiev, Ukraine
- United Kingdom (4):
  - Queen Elizabeth Hospital, Edgbaston, Birmingham
  - Leicester Royal Infirmary, Leicester, England
  - St. George's Hospital, London, England
  - Edinburgh Royal Infirmary, Edinburgh, Scotland